CLINICAL TRIAL: NCT00667524
Title: Eosinophilic Esophagitis: Influence of Esophageal Dilation on the Underlying Inflammation and Efficacy/Safety of the Procedure
Brief Title: Eosinophilic Esophagitis: Influence of Dilation on Dysphagia and Inflammation
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Dr Alain Schoepfer, Dpt of Gastroenerology, Bern University Hospital, Bern
Other Study IDs: KEK031_08
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Eosinophilic Esophagitis; Esophageal Stenosis; Esophageal Dilation; Esophageal Dilatation
Keywords: Eosinophilic Esophagitis; Dysphagia; Esophageal bougienage; Esophageal Dilation
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophageal Stenosis; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — formalin-fixed esophageal biopsies (blinded review of histology slides)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I

SUMMARY:
A database analysis and review of histological slides (retrospective) and a patient questionnaire analysis (prospective) will be conducted in Bern (Switzerland) to evaluate the efficacy and safety of esophageal dilation and its effect on the underlying eosinophilic inflammation in patients with Eosinophilic Esophagitis. This trial is investigator driven.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EE) is a chronic, increasingly recognized disease of the esophagus, clinico-pathologically characterized by a proton-pump-inhibitor resistant, dense esophageal eosinophilia in combination with esophagus-related symptoms. Patients suffer mainly from dysphagia, a feared long-term complication is the evolution of esophageal stenoses leading to food-bolus impaction that have to be removed endoscopically. Anti-inflammatory therapy with systemic or topical corticosteroids have shown to be efficacious in children as well as in adults. However, relapses occur in general soon after the cessation of this medication. In addition, several studies have demonstrated that in adults with active EE dilation is an alternative safe and efficacious therapeutic option. Surprisingly, the symptom-free period seems to be much longer after this procedure than after medical treatment. Today, the selection of these two procedures depends more on local practices than on evidence based data, because robust data are lacking. Furthermore, there are concerns regarding the risk of the dilation-procedure (possible esophageal perforations and major bleeding). Furthermore, it has not yet been assessed if dilation changes the underlying eosinophilic inflammation. If not, investigations should be performed to evaluate if long-term anti-eosinophilic therapy is able to change the natural course of the disease and reduce the stricturing complications.

ELIGIBILITY:
Inclusion criteria for retrospective Database analysis:

* Adult patients with - according to the database inclusion criteria - confirmed active EE, having

  1. Pre-dilational upper endoscopy (EGD) including histology and
  2. Dilation and
  3. Post-dilational EGD/Histo
* Definitions: Active EE is defined as

  1. Symptoms of dysphagia on almost each intake of solid food when off anti-inflammatory therapy or dietary restriction;
  2. Presence of an eosinophilic tissue infiltration with a peak cell density of >24 eosinophils per hpf x 400 on histology of esophageal biopsies.
* Inclusion criteria for additional, prospective, comprehensive histologic and immunologic
* Work-Up: "Comparable" time frame between baseline and post-dilational biopsy sampling

Exclusion criteria:

* Therapy with anti-eosinophilic medications 12 weeks prior to pre-dilational EGD and dilation respectively and between dilation and post-dilational EGD/Histo.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Eosinophilic Esophagitis referred to gastroenterologists in whole Switzerland working in private practice and in secondary and tertiary referral centers (Departments of Gastroenterology in hospitals)
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Assessment of eosinophilic esophageal infiltration before/after esophageal bougienage (without any anti-eosinophilic medication) | 3 months to 4 years

SECONDARY OUTCOMES:
Effect of dilation regarding dysphagia | 0 months to 4 years
Duration of a positive effect | 0 months to 4 years
Acceptance of dilation therapy by the patient | 0 months to 4 years after dilation therapy
Intensity of post-procedural pain | 1 day to 30 days after dilatation therapy
Duration of post-procedural pain | 1 day to 30 days after dilation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alain Schoepfer, Dr, Principal Investigator — Dpt of Gastroenterology, Bern University Hospital, Bern
Locations (1):
- Dpt of Gastroenterology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Background] Potter JW, Saeian K, Staff D, Massey BT, Komorowski RA, Shaker R, Hogan WJ. Eosinophilic esophagitis in adults: an emerging problem with unique esophageal features. Gastrointest Endosc. 2004 Mar;59(3):355-61. doi: 10.1016/s0016-5107(03)02713-5. PMID 14997131
- [Background] Ngo P, Furuta GT, Antonioli DA, Fox VL. Eosinophils in the esophagus--peptic or allergic eosinophilic esophagitis? Case series of three patients with esophageal eosinophilia. Am J Gastroenterol. 2006 Jul;101(7):1666-70. doi: 10.1111/j.1572-0241.2006.00562.x. PMID 16863575
- [Background] Straumann A, Spichtin HP, Grize L, Bucher KA, Beglinger C, Simon HU. Natural history of primary eosinophilic esophagitis: a follow-up of 30 adult patients for up to 11.5 years. Gastroenterology. 2003 Dec;125(6):1660-9. doi: 10.1053/j.gastro.2003.09.024. PMID 14724818
- [Background] Desai TK, Stecevic V, Chang CH, Goldstein NS, Badizadegan K, Furuta GT. Association of eosinophilic inflammation with esophageal food impaction in adults. Gastrointest Endosc. 2005 Jun;61(7):795-801. doi: 10.1016/s0016-5107(05)00313-5. PMID 15933677
- [Background] Baxi S, Gupta SK, Swigonski N, Fitzgerald JF. Clinical presentation of patients with eosinophilic inflammation of the esophagus. Gastrointest Endosc. 2006 Oct;64(4):473-8. doi: 10.1016/j.gie.2006.03.931. Epub 2006 Jul 26. PMID 16996334
- [Background] Konikoff MR, Noel RJ, Blanchard C, Kirby C, Jameson SC, Buckmeier BK, Akers R, Cohen MB, Collins MH, Assa'ad AH, Aceves SS, Putnam PE, Rothenberg ME. A randomized, double-blind, placebo-controlled trial of fluticasone propionate for pediatric eosinophilic esophagitis. Gastroenterology. 2006 Nov;131(5):1381-91. doi: 10.1053/j.gastro.2006.08.033. Epub 2006 Aug 16. PMID 17101314
- [Background] Remedios M, Campbell C, Jones DM, Kerlin P. Eosinophilic esophagitis in adults: clinical, endoscopic, histologic findings, and response to treatment with fluticasone propionate. Gastrointest Endosc. 2006 Jan;63(1):3-12. doi: 10.1016/j.gie.2005.07.049. PMID 16377308
- [Background] Schoepfer AM, Gschossmann J, Scheurer U, Seibold F, Straumann A. Esophageal strictures in adult eosinophilic esophagitis: dilation is an effective and safe alternative after failure of topical corticosteroids. Endoscopy. 2008 Feb;40(2):161-4. doi: 10.1055/s-2007-995345. PMID 18253909
- [Result] Schoepfer AM, Gonsalves N, Bussmann C, Conus S, Simon HU, Straumann A, Hirano I. Esophageal dilation in eosinophilic esophagitis: effectiveness, safety, and impact on the underlying inflammation. Am J Gastroenterol. 2010 May;105(5):1062-70. doi: 10.1038/ajg.2009.657. Epub 2009 Nov 24. PMID 19935783